CLINICAL TRIAL: NCT06443112
Title: Pregnancy Outcomes According To Cervical Cerclage Indications And Factors Affecting Pregnancy Duration And Outcomes: A 2-Year Comparison Of Patients Who Underwent History-Based, Ultrasound-Based, or Rescue Cerclage
Brief Title: Pregnancy Outcomes According to Cervical Cerclage Indications and Factors Affecting Pregnancy Duration and Outcomes
Acronym: CCERCIAFAO
Status: Completed | Type: Observational
Sponsor: Başakşehir Çam & Sakura City Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: BasaksehirCamveSakuraH
Record Dates: First submitted 2024-05-22; First posted 2024-06-05 (Actual); Last update posted 2024-06-05 (Actual); Status verified 2024-05

CONDITIONS: Cervical Incompetence (Complicating Pregnancy)
Keywords: cervical cerclage indications; cervical insufficiency; post-cerclage cervical length; Pregnancy outcomes
MeSH Terms: conditions — Uterine Cervical Incompetence; Pregnancy Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- history-indicated cerclage group (group1): Group 1 included patients with history-indicated cerclage, who had second-trimester pregnancy loss associated with painless cervical dilatation in the absence of labor or placental abruption, or previous cerclage due to painless cervical dilatation in the second trimester.
  Interventions: Procedure: transvaginal cervical cerclage by Mc Donald technique
- (Group 2) patients with ultrasound-indicated cerclage: Group 2 comprised patients with ultrasound-indicated cerclage, who had a history of spontaneous preterm birth before the 34th week previously and their cervical length was <25 mm before the 24th week of gestation in the current singleton pregnancy, or who had <10 mm cervical length in the current singleton pregnancy without history.
  Interventions: Procedure: transvaginal cervical cerclage by Mc Donald technique
- Group 3 consisted of patients undergoing rescue cerclage: Group 3 consisted of patients undergoing rescue cerclage, who had premature cervical dilatation and exposure of fetal membranes in the vagina, was detected in ultrasound or speculum examination of the cervix.
  Interventions: Procedure: transvaginal cervical cerclage by Mc Donald technique

INTERVENTIONS:
Procedure: transvaginal cervical cerclage by Mc Donald technique — In the McDonald operation, a suture is is inserted around the exo-cervix as high as possible to approximate to the level of the internal os and thereby prevent second-trimester abortion.

SUMMARY:
This study aimed to asses predictive factors associated with successful cervical cerclage and poor pregnancy outcomes in all indications.129 pregnant women who underwent cerclage at 12-25 weeks gestation in a perinatal medical center were included. The patients were divided into three subgroups for data analysis. Groups included patients with respectively history-indicated cerclage (group 1), ultrasound-indicated cerclage (group 2), and rescue cerclage (group 3). The investigators defined successful cerclage as postponing birth until after the 28th week of gestation and a 'good outcome' was defined as delivery beyond 34 completed weeks.Factors associated with successful cervical cerclage and perinatal outcomes after the procedure for all three groups were analyzed. The investigators also calculated post-cerclage the cervical length cut-off value required to predict if birth could be postponed until after the 28th week of gestation in women with cervical insufficiency.

DETAILED DESCRIPTION:
This study retrospectively reviewed data from pregnant women who underwent cerclage from July 2021 to July 2023 in Çam and Sakura City Hospital, which is a perinatal medical center in Istanbul, Turkey. The local ethics committee approved the study.

All procedures followed the relevant guidelines and regulations of the institutional ethics review board and the Declaration of Helsinki.

The patients were divided into three subgroups for data analysis. Group 1 included patients with history-indicated cerclage, who had second-trimester pregnancy loss associated with painless cervical dilatation in the absence of labor or placental abruption, or previous cerclage due to painless cervical dilatation in the second trimester. Group 2 comprised patients with ultrasound-indicated cerclage, who had a history of spontaneous preterm birth before the 34th week previously and their cervical length (CL) was <25 mm before the 24th week of gestation in the current singleton pregnancy, or who had <10 mm cervical length in the current singleton pregnancy without history. Group 3 consisted of patients undergoing rescue cerclage, who had premature cervical dilatation and exposure of fetal membranes in the vagina, was detected in ultrasound or speculum examination of the cervix. All cervical cerclage procedures were performed by a senior obstetrician using the McDonald technique with Mersilene tape or No:1 proline. The investigators collected the following data from medical records: maternal age at cervical cerclage, gravidity, parity, body mass index, history of a cervical cone biopsy, history of premature birth and cervical cerclage, procalcitonin level, C-reactive protein (CRP) level, gestational age at cerclage, pre-and post-cerclage CL, week of birth, pregnancy complications (preterm premature rupture of the membranes (PPROM), abruptio placenta, chorioamnionitis). The investigators defined successful cerclage as postponing birth until after the 28th week of gestation and a 'good outcome' was defined as delivery beyond 34 completed weeks. The indications and the pregnancy outcomes (miscarriage, gestational age at delivery, birth weight, prolongation of pregnancy, and rate of preterm birth before 34 weeks) of cervical cerclage were reviewed and the factors associated with successful cervical cerclage were analyzed.

Moreover, receiver operating characteristic (ROC) curves were used to calculate the pre-cerclage and post-cerclage CL cut-off value required to predict if birth could be postponed birth until after the 28th week of gestation in women with cervical insufficiency (CI). Thus, the investigators extracted significant factors for a successful cervical cerclage for long-term pregnancy sustenance in women with CI.

ELIGIBILITY:
Inclusion Criteria:

* Pregnants that underwent cervical cerclage between July 2021 and July 2023 with singleton pregnancies

Exclusion Criteria:

* Pregnant women without follow-up whose post-procedure data cannot be accessed
* Multiple pregnancies

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — pregnant women who underwent cerclage
Study Population: 18-45 aged Pregnant women who underwent cerclage at 12-25 weeks gestation from July 2021 to July 2023 in Çam and Sakura City Hospital, which is a perinatal medical center in Istanbul, Turkey.
Sampling Method: Probability Sample
Enrollment: 129 (Actual)
Dates: Start 2024-05-10 (Actual); Primary Completion 2024-05-10 (Actual); Study Completion 2024-05-10 (Actual)

PRIMARY OUTCOMES:
Latency from the time of cerclage procedure to delivery | time from cerclage procedure to birth
  Factors affecting time (time in days) elapsed from cerclage procedure to birth were evaluated
pre-cerclage and post-cerclage cervical length cut-off value required to predict if birth could be postponed birth until after the 28th week of gestation in women with cervical insufficiency. | time from diagnosis to birth
  receiver operating characteristic (ROC) curves were used to calculate the pre-cerclage and post-cerclage CL (length in centimeters) cut-off value required to predict if birth could be postponed birth until after the 28th week of gestation in women with CI. Thus, we extracted significant factors for a successful cervical cerclage for long-term pregnancy sustenance in women with CI.

CONTACTS AND LOCATIONS:
Overall Officials: Zeynep Kayaoglu yıldırım, MD, Study Director — Başakşehir Çam ve Sakura City Hospital; Elif Sagban Gedik, MD, Principal Investigator — Başakşehir Çam ve Sakura City Hospital
Locations (1):
- İstanbul Başakşehir Çam ve Sakura City Hospital, Istanbul, Basaksehir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Song RK, Cha HH, Shin MY, Choi SJ, Oh SY, Kim JH, Roh CR. Post-cerclage ultrasonographic cervical length can predict preterm delivery in elective cervical cerclage patients. Obstet Gynecol Sci. 2016 Jan;59(1):17-23. doi: 10.5468/ogs.2016.59.1.17. Epub 2016 Jan 15. PMID 26866031
- [Result] Chan LL, Leung TW, Lo TK, Lau WL, Leung WC. Indications for and pregnancy outcomes of cervical cerclage: 11-year comparison of patients undergoing history-indicated, ultrasound-indicated, or rescue cerclage. Hong Kong Med J. 2015 Aug;21(4):310-7. doi: 10.12809/hkmj144393. Epub 2015 Jul 17. PMID 26183455
- [Result] Cook JR, Chatfield S, Chandiramani M, Kindinger L, Cacciatore S, Sykes L, Teoh T, Shennan A, Terzidou V, Bennett PR. Cerclage position, cervical length and preterm delivery in women undergoing ultrasound indicated cervical cerclage: A retrospective cohort study. PLoS One. 2017 Jun 1;12(6):e0178072. doi: 10.1371/journal.pone.0178072. eCollection 2017. PMID 28570639

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-11-22): https://cdn.clinicaltrials.gov/large-docs/12/NCT06443112/Prot_SAP_000.pdf